CLINICAL TRIAL: NCT00720837
Title: Pilot Study Evaluating the Feasibility of Real-Time, Magnetic Resonance Thermal Imaging (MRTI) and Magnetic Resonance Imaging-Guided Laser Induced Thermal Therapy for Treatment of Metastatic Brain Tumors
Brief Title: Magnetic Resonance Temperature Imaging & Imaging-Guided Laser Induced Thermal Therapy for Treatment of Metastatic Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: BioTex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0610
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; Brain Cancer; MR-guided laser thermal ablation of brain tumors; Visualase® Thermal Therapy System; Magnetic Resonance Thermal Imaging; MRTI; Visualase Cooled Laser Application System; Laser Interstitial Thermal Therapy; LITT
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser Interstitial Thermal Therapy (Experimental): Laser Interstitial Thermal Therapy (LITT) - An intraoperative biopsy and placement of applicator for laser treatment. Treatment will last between 5 and 10 minutes.
  Interventions: Procedure: Visualase® Thermal Therapy System

INTERVENTIONS:
Procedure: Visualase® Thermal Therapy System — An intraoperative biopsy and placement of applicator for laser treatment. Treatment will last between 5 and 10 minutes.
  Other Names: Laser Interstitial Thermal Therapy (LITT)

SUMMARY:
The goal of this clinical research study is to learn about a new therapy device called the Visualase® Thermal Therapy System (a device that uses a laser to kill tumor cells and is guided using magnetic resonance thermal imaging [MRTI]). The Visualase® Thermal Therapy System is used to treat metastatic brain tumors. Researchers want to find out if it is possible to use this new device in patients with metastatic brain tumor(s), each measuring 3 centimeters (cm) or smaller. The safety of the device will also be studied.

DETAILED DESCRIPTION:
The Study Device and Process:

The Visualase® Thermal Therapy System combines 3 FDA-approved devices: the Visualase Cooled Laser Application System, which delivers the laser (energy) beams to the tumor tissue; the PhoTex 15 Diode Laser Series, which is the laser itself; and the Visualase ENVISION Workstation, which is the computer system that helps the surgeon plan and monitor your treatment.

The Visualase® Thermal Therapy System will be used in this study to give patients a type of therapy called Laser Interstitial Thermal Therapy (LITT). LITT uses laser light to heat and destroy the affected tissue; this is sometimes referred to as tissue ablation. In LITT, small fiber-optic applicators are placed directly into the tumor and heating is performed from the inside out, which may lead to the destruction of the tumor. During the heating process, MRTI can be used to watch the temperatures around the applicator to make sure that the tumor receives enough treatment and that the normal tissues around the tumor do not get too hot.

LITT is less invasive than an open surgical procedure. There are no radiation-related side effects, or limits on the number of times it can be repeated. Also, since the procedure is performed using the MRTI, doctors can find out right away how effective the therapy was by using special imaging sequences, which may also show any surviving tumor cells.

Screening:

Before you can enroll on this study, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed within 14 days before your treatment:

* Your medical history will be recorded, and you will be asked questions about any other treatment you have had for the metastatic brain tumor(s).
* You will have a complete physical exam.
* You will have a neurological exam. This will include an exam of the function of the nerves in your head, an exam of your visual fields, and tests of your reflexes, muscle strength, and senses.
* You will have an MRI scan of your brain within 30 days before LITT therapy.
* Women who are able to have children must have a negative urine pregnancy test within 48 hours (2 days) before treatment.

Study Treatment:

If you are found to be eligible to take part in the study, you will be scheduled for treatment of the brain tumor(s) using the Visualase® Thermal Therapy System.

You will be brought to a special operating room called the BrainSUITE®. The BrainSUITE® is a regular operating room that has a built-in MRI machine that can be used for taking pictures during the surgery. The imaging and procedure will be performed while you are under anesthesia (either deep sedation or fully "asleep").

A standard tumor biopsy will be performed. Then, using the same needle holder, the laser applicator will be placed within the tumor. MRI scans will be taken to make sure the applicator is placed properly. The biopsy and applicator placement will take about 1 hour.

After that, the laser treatment will be performed. At the same time, MRI scans will be taken during the procedure. The treatment will last between 5 and 10 minutes. After treatment, follow-up MRI scans will be taken, which may take 30-60 minutes longer. If any tumor tissue is left over, the laser may be moved slightly and a second treatment performed. Once completed, the needle will be removed, and your incision will be closed in the standard way.

If the tumor biopsy results reveal that the tumor has not come back, LITT will not be performed. Other treatment options which are available to you will be discussed with your doctor prior to the surgery.

Study Tests:

After the laser treatment, you will be observed in the hospital for 24 hours. While you are in the hospital, at about 1 day after treatment, you will have a physical and neurological exam, as well as a computed tomography (CT) scan of your brain (without using a contrast dye injected in the bloodstream) to make sure there were no problems with treatment. This is standard after any biopsy.

Follow-Up Testing:

You will be seen by your doctor for follow-up testing at about 1 week, 1 month, 3 months, and 6 months after your treatment. It will be very important for you to return to see your doctor at your scheduled visits, even if you are feeling fine. At the follow-up visits, your doctor will perform a complete physical and neurological exam. You will also have an MRI at all visits, starting with the 1-month visit.

This is an investigational study. Each part of the Visualase® Thermal Therapy System is FDA approved for use in delivering LITT to patients. Up to 22 patients will take part in this clinical research study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or family able and willing to give informed consent.
2. Subjects with metastatic cancer to the brain who have failed at least one conventional therapy (surgery, stereotactic radiosurgery, and/or whole brain radiotherapy). Failure is defined as local recurrence or failure of the previously treated lesion and will be determined by the treating surgeon based on a review of patient history and imaging.
3. Tumor size </= 3.0 cm in largest diameter.
4. MR imaging is not contraindicated for the patient
5. Lesion(s) are clearly defined on pre-therapy contrast enhanced MRI scans as determined by the treating surgeon.
6. Able and willing to attend all study visits.
7. Karnofsky Performance Scale score >/=70 for patients over the age of 15.
8. Lansky Play Scale>/=70 for patients 15 years of age or younger.

Exclusion Criteria:

1. Patients or family unwilling or unable to give written consent.
2. Patients who cannot physically fit in, or are too heavy for, the BrainSUITE® MRI scanner
3. Patients with contra-indications to MRI imaging, such as, but not limited to, pacemakers or defibrillators, non-compatible aneurysm clips, shrapnel, or other internal ferromagnetic objects
4. Known sensitivity to gadolinium-DTPA
5. Based on Treatment Planning Imaging (MR and/or CT) done on the day of treatment: -Brain edema and/or mass effect that causes midline shift or shift in wall of ventricle of more than 5 mm. -Lesions localized in the brain stem or the posterior fossa. -Lesions less than 5mm from primary branches of cerebral vessels, venous sinus, hypophysis or cranial nerves. -Evidence of recent (<2 weeks) hemorrhage.
6. Symptoms and signs of increased intracranial pressure
7. Medical issues which prohibit the patient from undergoing surgery (as determined by the treating surgeon, anesthesiologist, IMPAC clinic, referring physician).
8. Patients who are unable to received corticosteroids.
9. Positive pregnancy test for women of child-bearing age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Feasibility: Rate of technical success or failure to complete initial procedure with no associated major complications. | Safety: 30, 90, 180 day procedure-related morbidity and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weinberg, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org